CLINICAL TRIAL: NCT05295979
Title: Development of a Novel Chinese Medicine Formula for the Treatment of Psoriasis: A Randomized, Double-blinded, Placebo-controlled Trial
Brief Title: Chinese Medicine for Patients With Psoriasis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Lin Zhixiu, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Psoriasis study
Record Dates: First submitted 2022-02-24; First posted 2022-03-25 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inflammatory skin disease formula (ISDF) (Experimental): Subjects will receive ISDF granules (10.85g twice daily) for 12 weeks.
  Interventions: Drug: Inflammatory skin disease formula
- Placebo (Placebo Comparator): Subjects will receive placebo granules (10.85g twice daily) for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Inflammatory skin disease formula — ISDF granules (10.85g twice daily) for 12 weeks
  Other Names: ISDF
  Arms: Inflammatory skin disease formula (ISDF)
Drug: Placebo — Placebo granules (10.85g twice daily) for 12 weeks
  Arms: Placebo

SUMMARY:
Psoriasis is an inflammatory skin disease with huge negative impact on the quality of life of the patients, and has an overall prevalence of 2% to 3% in the general population. Plaques psoriasis is the most common type of the disease and presents red, well demarcated, and silvery plaques mainly localized in the umbilical and lumbosacral area as well as in the elbows, knees, and scalp.

Currently, pharmacological treatments such as retinoids, corticosteroids, vitamin D analogs and biologics remain the main options for most psoriasis patients. However, side effect and high cost barred many ordinary psoriasis patients.

A Chinese medicine formula "Inflammatory skin disease formula (ISDF)" was prescribed by Prof. Lin for many years and observed to be effective in relieving atopic dermatitis and psoriasis patients' clinical manifestations.

In this study, subjects with psoriasis will be randomized into treatment group of "ISDF" or placebo group for 12 weeks.

DETAILED DESCRIPTION:
Psoriasis is an inflammatory skin disease with huge negative impact on the quality of life of the patients, and has an overall prevalence of 2% to 3% in the general population. Plaques psoriasis is the most common type of the disease and presents red, well demarcated, and silvery plaques mainly localized in the umbilical and lumbosacral area as well as in the elbows, knees, and scalp. The major histological features of psoriasis include epidermal hyperplasia with aberrant keratinocyte differentiation, pronounced inflammatory cell infiltration and increased vascularization. Currently, pharmacological treatments such as retinoids, corticosteroids, and vitamin D analogs remain the main options for most psoriasis patients. However, the efficacy of conventional drugs is limited because of adverse side effects and the development of pharmacoresistance. Recently, biologics have become available for the treatment of acute and subacute plaque psoriasis with excellent response rate. However, the high costs involved with the biologics have barred many ordinary psoriasis patients from benefiting from this new class of anti-psoriatic medication. Natural products are valuable sources in novel drug development. Inflammatory skin disease formula (ISDF) is an empirical formula of the Principal Investigator (Prof. Zhi-Xiu Lin), a highly experienced Registered Chinese Medicine Practitioner and Chinese medicine dermatologist working at the School of Chinese Medicine, The Chinese University of Hong Kong. ISDF has been prescribed in clinic in Hong Kong for many years and observed to be effective in relieving atopic dermatitis and psoriasis patients' clinical manifestations. ISDF contains nine Chinese herbal medicines, including Rehmanniae Radix (Dihuang) 20.0 g, Paeoniae Radix Rubra (Chiyao) 10.0 g, Scutellariae Radix (Huangqin) 10.0 g, Phellodendri Cortex (Huangbai) 10.0 g, Forsythiae Fructus (Lianqiao) 12.0 g, Plantaginis Semen (Cheqianzi) 10.0 g, Vignae Semen (Chixiaodou) 10.0 g, Dictamni Cortex (Baixianpi) 10.0 g and Kochiae Fructus (Difuzi) 10.0 g. Among them, Rehmanniae Radix is frequently used for the treatment of psoriasis in Chinese medicine. Paeoniflorin, the major active ingredients of Paeoniae Radix Rubra, has been reported to inhibit imiquimod (IMQ)-induced psoriasis in mice by regulating Th17 cell response and cytokine secretion. Baicalin, the active components of Scutellariae Radix, was able to improve the psoriasis-like skin lesions induced by IMQ or 2,4-dinitrofluorobenzene (DNCB) in mice. Berberine, the main alkaloid of Phellodendri Cortex, could inhibit IMQ-induced psoriasis-like skin lesions and upregulation of CDC6 and p-STAT3 in mice.

Recent study demonstrated that ISDF (named SZF in the study) markedly decreased the epidermal thickening and infiltration of mast cells in the ears and dorsal skin of the DNCB-treated mice via inhibition of inflammation through inactivation of NF-κB p65 pathway. The ISDF was found to contain baicalin (4.92%, w/w), berberine (2.90%, w/w), paeoniflorin (0.26%, w/w) and phillyrin (0.10%, w/w). Recent preliminary data revealed that ISDF significantly improved the psoriatic-like symptoms and reduced the epidermal thickening in the dorsal skin of IMQ-stimulated mice via inhibition of the inflammation response. The results on its acute toxicity demonstrated that ISDF at up to the dose of 37.8 g/kg, which was the maximum tolerable dose of ISDF in mice, did not exert any overt toxicity. Based on these positive findings of pilot study, the investigators therefore hypothesize that ISDF is an effective herbal formula with anti-psoriatic effects. In Chinese medicine (CM) theory, psoriasis may be classified into different subtypes or "syndromes", including syndrome of wind-heat and blood heat, which is also known as blood heat syndrome or syndrome of wind-heat and blood dryness; syndrome of blood deficiency and wind-dryness; syndrome of blood stasis in the skin; and dampness-heat syndrome. Each of these syndromes represents a different pathogenesis in CM and corresponds to a different stage or manifestation of psoriasis. ISDF is composed of herbal medicines that can clear heat to cool the blood, clear heat and dry dampness, clear heat and drain dampness, disperse wind-heat, and is suitable for treating psoriasis with wind-heat, blood heat or dampness-heat. A randomized, double-blinded, placebo-controlled trial will be conducted to evaluate the efficacy of ISDF on psoriasis patients. Clinical evidence for the anti-psoriatic effects of ISDF, and is a necessary step towards developing this Chinese medicine formula into an anti-psoriatic pharmaceutical agent.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate chronic plaque psoriasis (PASI score 3 to 12).
* Willingness to give informed consent.

Exclusion Criteria:

* Pustular or generalized erythrodermic psoriasis.
* Psoriatic arthritis with syndrome of spleen-kidney yang deficiency according to Chinese medicine theory.
* Systemic therapy for psoriasis 6 months prior to baseline.
* Use topical medications for psoriasis 14 days prior to baseline such as retinoids, corticosteroids, vitamin D analogues, tazarotene and tacrolimus.
* Has taken any antibiotics, probiotics and prebiotics 30 days prior to baseline.
* UV light therapy 30 days prior to baseline.
* Clinically significant laboratory abnormality in blood, liver or renal functions (≥1.5 times the upper limit of reference range).
* History of allergy to Chinese herbs.
* Unwillingness to comply with study protocol.
* Any other condition that in the opinion of the investigators could compromise the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Psoriasis Area and Severity Index (PASI) | Week 12
  The change in Psoriasis Area and Severity Index (PASI) score will be assessed. PASI scores include area involved, erythema, induration and scaling. It will be scored on a scale of 0 to 4 (0, meaning none; 1, mild; 2, moderate; 3, severe; and 4, very severe). It will be performed by 2 blinded assessors who have been trained. Four main areas were assessed for calculation of the PASI scores: the head, the trunk, the upper extremities, and the lower extremities, corresponding to 10%,20%,30%, and 40% of the total body area, respectively. The maximum score for PASI is 72.
Static Physician Global Assessment score (sPGA) | Week 12
  Participants are requested to expose their skin thoroughly before the photographs are taken at each visit. The sPGA is an investigator-rated assessment of overall disease severity to be evaluated on a 5-point scale, where 0=clear and 4=severe. The severity of erythema, scaling, and plaque are considered for assessment. It will be performed by 2 blinded assessors who have received training.

SECONDARY OUTCOMES:
Psoriasis Area and Severity Index (PASI) | Week 6
  The change in Psoriasis Area and Severity Index (PASI) score will be assessed. PASI scores include area involved, erythema, induration and scaling. It will be scored on a scale of 0 to 4 (0, meaning none; 1, mild; 2, moderate; 3, severe; and 4, very severe). It will be performed by 2 blinded assessors who have been trained. Four main areas were assessed for calculation of the PASI scores: the head, the upper extremities, the trunk, and the lower extremities, corresponding to 10%,20%,30%, and 40% of the total body area, respectively. The maximum score for PASI is 72.
Psoriasis Area and Severity Index (PASI) | Week 18
  The change in Psoriasis Area and Severity Index (PASI) score will be assessed. PASI scores include area involved, erythema, induration and scaling. It will be scored on a scale of 0 to 4 (0, meaning none; 1, mild; 2, moderate; 3, severe; and 4, very severe). It will be performed by 2 blinded assessors who have been trained. Four main areas were assessed for calculation of the PASI scores: the head, the upper extremities, the trunk, and the lower extremities, corresponding to 10%,20%,30%, and 40% of the total body area, respectively. The maximum score for PASI is 72.
Static Physician Global Assessment score (sPGA) | Week 6
  Participants are requested to expose their skin thoroughly before the photographs are taken at each visit. The sPGA is an investigator-rated assessment of overall disease severity to be evaluated on a 5-point scale, where 0=clear and 4=severe. The severity of erythema, scaling, and plaque are considered for assessment. It will be performed by 2 blinded assessors who have received training.
Static Physician Global Assessment score (sPGA) | Week 18
  Participants are requested to expose their skin thoroughly before the photographs are taken at each visit. The sPGA is an investigator-rated assessment of overall disease severity to be evaluated on a 5-point scale, where 0=clear and 4=severe. The severity of erythema, scaling, and plaque are considered for assessment. It will be performed by 2 blinded assessors who have received training.
Impact of Psoriasis Questionnaire (IPSO) | Week 12
  The change in Impact of Psoriasis Questionnaire (IPSO) score will be assessed. IPSO is a validated 16-item psoriasis-specific instrument for quality of life of psoriasis patients. The IPSO is intended predominantly to assess the psychosocial impact of psoriasis on patient's lives. The IPSO uses an ordinal rating scale, with responses of 'none', 'some', 'moderately', 'quite a bit' and 'extremely' scored 1, 2, 3, 4 and 5, respectively. The scores for item 4 were reversed. The higher the summed score, the greater the impact experienced due to psoriasis.
Short Form 36 survey (SF36) | Week 12
  The change in the score of quality of life using Short Form 36 survey (SF36) will be assessed. SF36 is generic instrument to measure general health status that is complementary to those derived from dermatological questionnaires. It will be used to assess the patient's health status using 8 different dimensions including vitality, physical functioning, bodily pain, general health perceptions, role limitations due to physical health, role limitations due to emotional health, social role functioning and mental health. The possible score ranges from 0 to 100 points whereby 0 points represent the greatest possible limitation of health, while 100 points represent the absence of health restrictions.
Use of rescue therapy | Up to Week 18
  The frequent use of rescue therapy during study period
Adverse events | Up to Week 18
  Adverse events related to study treatment
Serum markers (IL-17A, IL-22, IL-23, CRP and BD-2) | Week 12
  The changes in levels of serum markers [IL-17A, IL-22, IL-23, C-reactive protein (CRP) and Beta-Defensin 2 (BD2)].
Oral and Gut microbiota composition in saliva and stools | Week 12
  The changes in the oral and gut microbiota composition in saliva and stools
Psoriasis Itch Visual Analog Scale (Itch VAS) | Week 12
  Psoriasis itch VAS is a validated tool to assess treatment benefit of plaque psoriasis. It was developed to measure itch intensity within the last 24 hours. A horizontal line with a length of 100mm is to be used to represented the range of itch intensity from 0 (no itch at all) to 100 (worst itch you can imagine). Subjects rated the maximal intensity of itch during the previous 24 hours by putting a vertical mark through the horizontal line at the the spot he/she felt best reflected their maximal itch intensity.
Psoriasis-involved body surface area (BSA) | Week 6
  BSA represents the affected skin surface. It is an objective measure of psoriasis severity. The head, the upper extremities, the trunk, and the lower extremities, corresponding to 10%,20%,30%, and 40% of the total body area, respectively. The range of BSA is 0-100. It will be performed by 2 blinded assessors who have received training.
Psoriasis-involved body surface area (BSA) | Week 12
  BSA represents the affected skin surface. It is an objective measure of psoriasis severity. The head, the upper extremities, the trunk, and the lower extremities, corresponding to 10%,20%,30%, and 40% of the total body area, respectively. The range of BSA is 0-100. It will be performed by 2 blinded assessors who have received training.
Psoriasis-involved body surface area (BSA) | Week 18
  BSA represents the affected skin surface. It is an objective measure of psoriasis severity. The head, the upper extremities, the trunk, and the lower extremities, corresponding to 10%,20%,30%, and 40% of the total body area, respectively. The range of BSA is 0-100. It will be performed by 2 blinded assessors who have received training.

CONTACTS AND LOCATIONS:
Overall Officials: Zhixiu Lin, PhD, Principal Investigator — Hong Kong Institute of Integrative Medicine
Locations (1):
- Hong Kong Institute of Integrative Medicine, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No